CLINICAL TRIAL: NCT00625300
Title: Efficacy and Safety Study:The Influence of Repetitive Transcranial Stimulation (r-TMS) Treatment on Motor and Cognitive Measurements in Patients With Parkinson's Disease
Brief Title: Repetitive Transcranial Stimulation (r-TMS) Treatment for Patients With Parkinson's Disease
Acronym: r-TMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Dr. Oren Cohen- Principal investigator, Shema Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-08-4726-OC-CTIL
Record Dates: First submitted 2008-02-13; First posted 2008-02-28 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Parkinson's Disease
Keywords: repetitive transcranial stimulation; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Active treatment group: each patient will be given 3 treatment sessions per week for 4 weeks (a total of 12 sessions). Each session is 20 minutes long and will be consisted of 20Hz stimulation trains (active) over the motor cortex and the prefrontal cortex.
  Interventions: Device: repetitive transcranial stimulation (r-TMS)
- Placebo (Sham Comparator): Sham treatment group: each patient will be given 3 treatment sessions per week for 4 weeks (a total of 12 sessions). Each session is 20 minutes long and will be consisted of 20Hz stimulation trains (sham) over the motor cortex and the prefrontal cortex.
  Interventions: Device: Repetitive transcranial stimulation

INTERVENTIONS:
Device: repetitive transcranial stimulation (r-TMS) — Each patient will be given 3 treatment sessions per week for 4 weeks (a total of 12 sessions). Each session is 20 minutes long and will be consisted of 20Hz stimulation trains (active) over the motor cortex and the prefrontal cortex.
  Arms: 1
Device: Repetitive transcranial stimulation — Sham treatment group: each patient will be given 3 treatment sessions per week for 4 weeks (a total of 12 sessions). Each session is 20 minutes long and will be consisted of sham stimulation trains over the motor cortex and the prefrontal cortex.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the effects of deep rTMS using the novel H-coil on the motor, affective and cognitive deficits in patients with Parkinson's disease (PD) and to establish its safety in this population.

DETAILED DESCRIPTION:
Study rational:We anticipate that reaching deeper brain layers and larger volume of activation with the novel H-coil may induce significantly better therapeutic effects in patients with PD and will pave the way for establishing a novel and effective treatment for this disorder.

Design:A prospective, double blind sham-controled study. No. of centers:1 One: Tel-Hashomer Medical Center, affiliated to Sackler school of Medicine, Tel -Aviv University, Israel.

Study Population:Forty patients with idiopathic PD, Hoehn and Yahr stages II to IV, on stable antiparkinsonian therapy, with partial response.

Study Duration:Two years

ELIGIBILITY:
Inclusion Criteria:

* PD patients aged 40 years or older, diagnosed as idiopathic PD according to the UK Brain Bank criteria, with Hoehn & Yahr stages II - IV while "off". Participants on antidepressants should be at least 2 months on stable therapy.

Exclusion Criteria:

* Patients who have concomitant epilepsy, a history of seizure or heat convulsion or history of epilepsy in first degree relative.
* Patients on neuroleptics.
* Patients with dementia or any unstable medical disorder.
* History or current hypertension.
* History of head injury or neurosurgical interventions.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps.
* History of migraine or frequent or severe headaches.
* History of hearing loss.
* The presence of cochlear implants
* History of drug abuse or alcoholism.
* Pregnancy or not using a reliable method of birth control.
* Participation in current clinical study or clinical study within 30 days prior to this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson Disease Rating Scale (UPDRS)(Motor Part) | 10-90 days

SECONDARY OUTCOMES:
Clinical Global Impression of Severity (CGIS) | 10-90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel